CLINICAL TRIAL: NCT04395313
Title: Gender Discrimination Against Female Surgeons May Pass Unrecognized: A Study in a Lower-Middle-Income Country
Brief Title: Gender Discrimination Against Female Surgeons A Study in a Lower-Middle-Income Country
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, hina inam, Instructor, Aga Khan University
Other Study IDs: Gender discrimination
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Gender Issues
MeSH Terms: conditions — Sexism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention carried out — no intervention was done

SUMMARY:
our study explores how GD is perceived and reported by surgeons in Pakistan.

DETAILED DESCRIPTION:
Due to an increasing spotlight, gender discrimination (GD) is identified and reported in many aspects of surgical training and practice in the developed world 1, 2. In contrast, lower-middle-income countries like Pakistan lack awareness and strategies to counteract GD, which manifests as a lack of females in leadership and academic positions, and pay inequities. GD often occurs insidiously, as a result of complex interplay between societal norms, gender stereotypes and learned behaviors. Thus, our study identifies how GD is perceived and reported by surgeons in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* all consultants
* fellows
* instructors
* medical officers
* residents working in the Department of Surgery

Exclusion Criteria:

* all consultants
* fellows
* instructors
* medical officers
* residents not working in the Department of Surgery

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: all consultants
  * fellows
  * instructors
  * medical officers
  * residents working in the Department of Surgery
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
gender bias | 2 months
  Gender bias faced by female surgeons

SECONDARY OUTCOMES:
experience of gender discrimination | 2 months
  as in by whom were they gender discriminated

OTHER OUTCOMES:
impact | 2 months
  what was the impact of the gender discrimination

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Stadium Road, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: here you can email us and contact us to get details — https://mail.aku.edu/owa